CLINICAL TRIAL: NCT01823861
Title: Mobile Technology for Improved Family Planning
Acronym: MOTIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marie Stopes International (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MarieStopes
Record Dates: First submitted 2013-03-30; First posted 2013-04-04 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Contraception; Post-abortion Family Planning; mHealth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobile phone-based intervention (Experimental): Standard care plus automated voice message to support post-abortion contraception use every two weeks for total of three months and direct follow up phone call by family planning counsellor depending on response to voice message.
  Interventions: Behavioral: Mobile phone-based intervention
- Standard care (No Intervention): Face-to-face post-abortion family planning (PAFP) counselling, follow-up at one or two weeks, clinic phone number, existing 'Hotline' phone number.

INTERVENTIONS:
Behavioral: Mobile phone-based intervention — Automated voice message to support post-abortion contraception use every two weeks for total of three months. Direct follow up phone call by family planning counsellor depending on response to voice message.
  Arms: Mobile phone-based intervention

SUMMARY:
An individual randomised controlled trial (RCT) to evaluate the effectiveness of a voice-based mobile phone health (mHealth) intervention to support post-abortion family planning (PAFP) at four Marie Stopes International clinics in Cambodia.

The study seeks to address the research question: does a PAFP mHealth intervention increase use of contraception in Cambodia? STUDY RESULTS: http://www.who.int/bulletin/online_first/en/

ELIGIBILITY:
Inclusion Criteria:

* Client attending for abortion
* Client does not want to have a child at the current time
* Client aged 18 or over
* Client owns a mobile phone
* Client willing to receive simple voice messages relating to contraception from Marie Stopes in Khmer language

Exclusion Criteria:

* Not meeting inclusion criteria
* Declined to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Marie Stopes International, Phnom Penh, Cambodia

REFERENCES:
- [Result] Smith C, Ngo TD, Gold J, Edwards P, Vannak U, Sokhey L, Machiyama K, Slaymaker E, Warnock R, McCarthy O, Free C. Effect of a mobile phone-based intervention on post-abortion contraception: a randomized controlled trial in Cambodia. Bull World Health Organ. 2015 Dec 1;93(12):842-50A. doi: 10.2471/BLT.15.160267. Epub 2015 Oct 15. PMID 26668436
- [Derived] Hill J, McGinn J, Cairns J, Free C, Smith C. A Mobile Phone-Based Support Intervention to Increase Use of Postabortion Family Planning in Cambodia: Cost-Effectiveness Evaluation. JMIR Mhealth Uhealth. 2020 Feb 25;8(2):e16276. doi: 10.2196/16276. PMID 32130166
- [Derived] Smith C, Edwards P, Free C. Assessing the validity and reliability of self-report data on contraception use in the MObile Technology for Improved Family Planning (MOTIF) randomised controlled trial. Reprod Health. 2018 Mar 15;15(1):50. doi: 10.1186/s12978-018-0494-7. PMID 29544520
- [Derived] Smith C, Jarvis C, Free C. Assessing loss to follow-up in the MObile Technology for Improved Family Planning (MOTIF) randomised controlled trial. Trials. 2017 Dec 1;18(1):577. doi: 10.1186/s13063-017-2316-6. PMID 29191231
- [Derived] Smith C, Ngo TD, Edwards P, Free C. MObile Technology for Improved Family Planning: update to randomised controlled trial protocol. Trials. 2014 Nov 12;15:440. doi: 10.1186/1745-6215-15-440. PMID 25388660
- [Derived] Smith C, Vannak U, Sokhey L, Ngo TD, Gold J, Khut K, Edwards P, Rathavy T, Free C. MObile Technology for Improved Family Planning Services (MOTIF): study protocol for a randomised controlled trial. Trials. 2013 Dec 12;14:427. doi: 10.1186/1745-6215-14-427. PMID 24330763

RESULTS

PARTICIPANT FLOW:
Period: 4 Month Follow up
Arm/Group | Mobile Phone-based Intervention | Standard Care
Started | 249 | 251
Completed | 211 | 220
Not Completed | 38 | 31
Period: 12 Month Follow up
Arm/Group | Mobile Phone-based Intervention | Standard Care
Started | 211 | 220
Completed | 169 | 159
Not Completed | 42 | 61

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Phone-based Intervention | Standard Care | Total
Number analyzed (Participants) | 249 | 251 | 500
Age, Customized [Count of Participants; unit: Participants]
  <25 | 88 | 69 | 157
  ≥25 | 161 | 182 | 343
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 249 | 251 | 500
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Use of a Effective Contraceptive Method at Four-months Post-abortion
Description: Self-reported use of pill, coil, implant or injection for all participants. Objective measurement of contraceptive use for participants from one clinic.
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Mobile Phone-based Intervention | Standard Care
Number analyzed (Participants) | 211 | 220
participants | 135 | 101

2. Secondary Outcome: Pregnancy
Time Frame: 4 months
Reporting Status: Not Posted

3. Secondary Outcome: Repeat Abortion
Time Frame: 4 months
Reporting Status: Not Posted

4. Secondary Outcome: Contraceptive Discontinuation
Time Frame: 4 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Mobile Phone-based Intervention | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/249 | 0/251
Other Adverse Events (participants affected / at risk) | 0/249 | 0/251

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No